CLINICAL TRIAL: NCT05968664
Title: Novel Stimulation Patterns to Improve the Effectiveness of Spinal Cord Stimulation
Acronym: DYNAMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ashwin Viswanathan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Ashwin Viswanathan, Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H-49405; 4UH3NS121563-02 (NIH)
Record Dates: First submitted 2023-07-07; First posted 2023-08-01 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-06

CONDITIONS: Chronic Pain; Pain, Neuropathic; Neuropathic Pain
Keywords: Chronic pain; Spinal Cord Stimulation; Spinal cord; Neuropathy
MeSH Terms: conditions — Chronic Pain; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Time Invariant Pulse(TIP) Stimulation (Active Comparator): The control arm for this study will be the Time Invariant Pulse stimulation which is used in standard of care Spinal Cord Stimulation therapy. TIP tonic stimulation is delivered with fixed amplitude, pulse width, and frequency parameters.
  Interventions: Device: Spinal Cord Stimulator
- Time Variant Pulse (TVP) Stimulation (Experimental): The time variant pulse (TVP) stimulation will serve as the experimental arm for this study. There are two ways of delivering TVP stimulation to the spinal cord. TVP stimulation can either vary in intensity or it can vary rate, referred to as intensity-modulated TVP or rate-modulated TVP, respectively.
  Interventions: Device: Spinal Cord Stimulator

INTERVENTIONS:
Device: Spinal Cord Stimulator — Spinal Cord Stimulator modified to deliver Time Variant Pulse (TVP) stimulation.
  Arms: Time Variant Pulse (TVP) Stimulation
Device: Spinal Cord Stimulator — Spinal Cord Stimulator to deliver standard of care Time Invariant Pulse (TIP) stimulation.
  Arms: Time Invariant Pulse(TIP) Stimulation

SUMMARY:
The goal of this study is to compare pain outcomes achieved by spinal cord stimulation (SCS) using time varying stimulation patterns with pain outcomes achieved by current standard of care SCS.

DETAILED DESCRIPTION:
The researchers will conduct a traditional exploratory feasibility study using an investigational device to compare the clinical outcomes using time varying pulse (TVP) waveforms against time-invariant pulse (TIP) waveforms using both paresthesia and paresthesia-free SCS therapies. The therapy longevity of TVPs and TIPS will also be evaluated by tracking therapy efficacy through a long-term follow-up phase, using multiple pain assessments and at-home digital data collection.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Age ≥ 22
* Chronic pain of the trunk and/or limbs for at least 6 months
* Baseline average daily overall pain score of >60 (on a scale of 0-100mm) on the Visual Analog Scale related to pain of the back and/or limbs
* Failed ≥3 medically supervised treatments (i.e. pain medications, physical therapy, facet joint/medial branch nerve blocks, acupuncture), and treatment with >2 classes of medications
* Stable pain-related medication regimen 4 weeks prior to the trial. Patients will be asked to not increase or add pain-related medication during the study period
* No back surgery within 6 months prior to Screening
* Consumed an average total daily morphine equivalent of ≤200 mg during the 30 days prior to Screening.
* Baseline Oswestry Disability Index score ≥40 and ≤80
* Eligible candidate for SCS from a psychological and psychiatric standpoint as determined within 180 days prior to Baseline Visit, per site's routine screening process
* Able to independently read and complete all questionnaires and assessments provided in English
* Female candidates of child-bearing potential agree to use contraception during the study period
* Deemed to be a good candidate for spinal cord stimulation by the PI, and a board certified pain management physician
* Willing to cooperate with study requirements

Exclusion Criteria:

* Patient exhibits catastrophization based on physician evaluation (e.g., average overall daily pain intensity of 100 on a 0-100mm visual analog scale, every day during the 7 days prior to Screening, based on patient recall
* Pain originating from peripheral vascular disease
* Active treatment for cancer in past 6 months
* Involved in disability litigation
* High surgical risk including documented history of allergic response to titanium or silicone, current systemic infection, or local infection in close proximity to anticipated surgical field
* Body mass index ≥ 45 at Screening
* Terminal illness with anticipated survival < 12 months
* Participant is immunocompromised
* Significant cognitive impairment at Screening that, in the opinion of the Investigator, would reasonably be expected to impair the study candidate's ability to participate in the study
* Participating (or intends to participate) in another drug or device clinical trial that may influence the data that will be collected for this study
* Previous spinal cord stimulation trial/implant or is already implanted with an active implantable device(s) (e.g. drug pump, implantable pulse generator)
* A pregnant female or a female of childbearing potential planning to get pregnant during the course of the study
* Plan to receive any massage or manipulation directly over the leads or by the anticipated location of the IPG or treatments that involve sudden jerking motions of the torso at any
* Existing medical condition that is likely to require the use of diathermy
* Any injury or medical/psychological condition that might be significantly exacerbated by the implant surgery or the presence of an implantable stimulator or otherwise compromise subject safety
* Unable to operate the study devices including wrist-worn biosensor and mobile app
* Documented history of substance abuse or dependency in the 6 months prior to baseline

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in Patient responder rate | Patient responder rate will be measured from the baseline and during three experimental stimulation periods which are 8±3 weeks each.
  The primary endpoint for this trial will be a comparison of the percentage of patients achieving at least a 50% reduction in pain during the TIP stimulation block with the percentage of patients achieving at least a 50% reduction in pain during either TVP stimulation block.

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Viswanathan, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code